CLINICAL TRIAL: NCT05179083
Title: Regenerating the Adult Human Brain Through Exercise
Brief Title: Exercise for Brain Regeneration in Epilepsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jonathan Russin, Assistant Professor of Clinical Neurological Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: APP-21-04349
Record Dates: First submitted 2021-11-30; First posted 2022-01-05 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Temporal Lobe Epilepsy
Keywords: Exercise; Neurogenesis; Mesial temporal lobe epilepsy; Regeneration; Cognition; Electrophysiology
MeSH Terms: conditions — Epilepsy, Temporal Lobe; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-impact Exercise (Experimental)
  Interventions: Other: High-Impact Aerobic Exercise
- Low-impact Exercise (Active Comparator)
  Interventions: Other: Low-Impact Aerobic Exercise

INTERVENTIONS:
Other: High-Impact Aerobic Exercise — Participants will be submitted to a 12-week high-impact aerobic exercise program using a recliner bike with three sessions per week. The exercise protocol takes 45 minutes per session and consists of five minutes of warm-up, 30 minutes of cycling with progressive increase in intensity until the target heart rate (80% of maximum) is reached, followed by 10 minutes of cool down.
  Arms: High-impact Exercise
Other: Low-Impact Aerobic Exercise — Participants will be submitted to a 12-week low-impact aerobic exercise program using a recliner bike with three sessions per week. The exercise protocol takes 45 minutes per session and consists of five minutes of warm-up, 30 minutes of cycling with progressive increase in intensity until the target heart rate (40% of maximum) is reached, followed by 10 minutes of cool down.
  Arms: Low-impact Exercise

SUMMARY:
Nearly 100 million Americans are affected by neurological disorders with an overall cost above $765 billion for the more prevalent conditions. Given this significant burden, effective treatments to prevent dementia and new disease modifying therapies are urgently needed.

Regeneration of lost neurons with new ones (i.e., neurogenesis) is compromised at early stages of dementia and in part correlates with cognitive impairment in Alzheimer's disease. Boosting the neurogenesis delays the cognitive impairment in animal models of dementia and has been proven beneficial in improving the memory in rodent studies.

Aerobic exercise is the most potent known stimulator of neurogenesis in animal models. A crucial next step is to translate endogenous regenerative strategies to people. The purpose of this study is to demonstrate the feasibility and investigate the effects of an exercise program on neurogenesis and cognitive improvement in epilepsy patients.

DETAILED DESCRIPTION:
Neurogenesis studies in healthy and dementia patients have only been performed on postmortem tissue, which prevents investigation of treatment outcomes. Patients with mesial temporal lobe epilepsy (MTLE) typically do not respond to medications and uniquely among related dementia disorders undergo corrective surgical treatment, providing a unique opportunity to study the value of regenerative interventions on hippocampal electrophysiology and neurogenesis. Using this unique approach, this study will investigate the neurogenesis and cognitive improvement in epilepsy patients.

Ten people with MTLE who are recommended for surgical treatment as part of their standard care will be enrolled and randomly assigned to High Impact (n=5) and Low Impact (n=5) exercise groups. The duration of exercise programs will be 12 weeks and study arms will undergo the same protocol except for the target heart rate which will be higher in the High-Impact group. Exercise will be performed at home using a recliner bike under the supervision of caregiver and study personnel. Participants will undergo cognitive, exercise and clinical assessment at baseline and after completing the three-month exercise therapy; then surgically resected tissue will be analyzed for regeneration and epileptiform activity. The investigators will assess whether exercise would yield clinical benefits in terms of seizure frequency/intensity or cognitive ability, and whether the ability of the adult human brain to self-repair can be enhanced. It is hypothesized that the proposed exercise regimen is feasible and will improve the neurogenesis levels and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Medically resistant mesial temporal lobe epilepsy
* Candidacy for standard or selective temporal lobectomy

Exclusion Criteria:

* Age of older than 65 years
* Pregnancy
* Physical disabilities or medical conditions preventing from participation in exercise program
* Inability to receive exercise equipment at home
* Cognitive/developmental disabilities restricting the participation in exercise program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to exercise and assessments | Through study completion, an average of 6 months
  Number of completed exercise and assessment sessions

SECONDARY OUTCOMES:
Neurogenesis | 13 weeks after first exercise session
  Number of new neurons per mm3 in surgically resected tissue after cell culture
Rey Auditory Verbal Learning Test (RAVLT) - Trial V | Baseline and 12 weeks after first exercise session
  The Rey Auditory Verbal Learning Test (RAVLT) is a validated test evaluating verbal learning and memory. In this test, lists of words are read to the participants in consecutive trials. Trial V is the 5th attempt at recalling the first list of words.
Rey Auditory Verbal Learning Test (RAVLT) - Summary score | Baseline and 12 weeks after first exercise session
  The Rey Auditory Verbal Learning Test (RAVLT) is a validated test evaluating verbal learning and memory. In this test, lists of words are read to the participants in consecutive trials. Summary score is the sum of number of words learned over five learning trials.
WAIS-IV - Matrix Reasoning | Baseline and 12 weeks after first exercise session
  Wechsler Adult Intelligence Scale Fourth Edition (WAIS-IV) is a validated test of cognitive ability and intelligence. Matrix reasoning is among the tasks included in WAIS-IV which is used to assess non-verbal abstract problem solving and inductive reasoning.
Rey Complex Figure Test (RCFT) | Baseline and 12 weeks after first exercise session
  Rey Complex Figure Test (RCFT) is a standardized test of visuospatial memory. Performance will be scored based on the delayed recall trial of the RCFT.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Russin, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California Department of Neurosurgery, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gooch CL, Pracht E, Borenstein AR. The burden of neurological disease in the United States: A summary report and call to action. Ann Neurol. 2017 Apr;81(4):479-484. doi: 10.1002/ana.24897. No abstract available. PMID 28198092